CLINICAL TRIAL: NCT00204815
Title: Bone Mineral Density in Pediatric Epilepsy: AED-Specific and Duration of Treatment-Specific Effects
Brief Title: Bone Mineral Density in Pediatric Epilepsy
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 2004-0015
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
What are the effects of the currently used AEDs on bone mineralization in children and adolescents between the ages of 8 to 18? This is a pilot observational study using DEXA scans to measure bone mineral density in 100 patients The primary objective is to collect preliminary data on bone mineral density, body weight, dietary calcium intake, and activity level.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of generalized or partial seizures with or without generalization or a diagnosis of generalized seizures as defined in the International League Against Epilepsy

Exclusion Criteria:

* steroid use
* chronic disease other than epilepsy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric subjects with generalized or partial seizures
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2005-01; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj Sheth, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States